CLINICAL TRIAL: NCT07138001
Title: A Randomized, Controlled, Open-label, Multicenter Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of KH617 in Combination With Temozolomide Versus Investigator's Choice Treatment or KH617 Monotherapy for Recurrent Glioblastoma
Brief Title: Phase 2 Clinical Trial of KH617
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Honghe Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KH617-30201
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Platinum; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KH617+TMZ (Experimental): KH617： 33mg/kg intravenous infusion, every 4 weeks as one cycle.
  TMZ（5/28）：150~200mg/m2/d, oral, every 4 weeks as one cycle.
  Interventions: Combination Product: KH617+TMZ
- KH617 (Experimental): KH617： 33mg/kg intravenous infusion, every 4 weeks as one cycle.
  Interventions: Drug: KH617
- TPC: TMZ or Platinum (cisplatin or carboplatin)+VP-16 (Active Comparator): TMZ（7/7）： 100-150 mg/m2/d，oral, alternating weekly,every 4 weeks as one cycle.
  Platinum (cisplatin or carboplatin)+VP-16： Cisplatin for injection 80-100mg/m2, divided into 3 days, the dose depends on tolerability, every 4 weeks as one cycle; carboplatin injection 75-100mg/m2/d, continuously administered for 3 days, the dose depends on tolerability, every 4 weeks as one cycle; etoposide injection 100mg/m2/d, continuously administered for 3 days, every 4 weeks as one cycle.
  Interventions: Drug: TPC: TMZ or Platinum (cisplatin or carboplatin)+VP-16

INTERVENTIONS:
Combination Product: KH617+TMZ — use KH617 and TMZ(5/28) as Combination Product.
  Arms: KH617+TMZ
Drug: KH617 — Single Clinical trial investigational drug
  Arms: KH617
Drug: TPC: TMZ or Platinum (cisplatin or carboplatin)+VP-16 — Comparator product, Two treatment options for physicians and subjects to choose from:
  1. use TMZ(7/7)
  2. Use Platinum (cisplatin or carboplatin)+VP-16
  Arms: TPC: TMZ or Platinum (cisplatin or carboplatin)+VP-16

SUMMARY:
To evaluate the efficacy and safety of KH617 for injection in combination with temozolomide versus investigator's choice therapy or KH617 monotherapy for recurrent glioblastoma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female,age≥18 years old.
2. Life expectancy of at least 3 months.
3. Glioblastoma confirmed by histopathology.
4. Glioblastoma that recurred for the first time after failure of standard treatment.
5. Patient has at least one measurable lesion by iRANO.
6. MGMT promoter is unmethylated.
7. KPS≥ 60.
8. Adequate organ and bone marrow reserve function.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women or men who are planning to have children.
2. Patients who have received the following treatments before enrollment should be excluded:

   1. Patients who have received surgery, chemotherapy, targeted and immune drug therapy, iodine internal radiation, or radiotherapy within 4 weeks or 5 half-lives (whichever is shorter) before enrollment or who plan to receive radiotherapy during the trial.
   2. Patients who had undergone intracranial lesion biopsy within 7 days before enrollment.
   3. Received other clinical research drugs or treatments within 4 weeks before enrollment.
   4. Received treatment with traditional Chinese medicine or Chinese patent medicine with anti-tumor effects within 1 week before enrollment.
3. History of central nervous system hemorrhage/infarction, such as ischemic/hemorrhagic stroke, within 6 months before enrollment.
4. Known history of unstable angina, myocardial infarction, or congestive heart failure within the past 6 months or clinically significant arrhythmia requiring antiarrhythmic therapy.
5. Poorly controlled high blood pressure or diabetes.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites.
7. Patients at risk for active autoimmune disease or those with a history of autoimmune disease that may involve the central nervous system.
8. Pulmonary disease defined as grade ≥3 according to NCI-CTCAE v5.0.
9. Significant active bleeding within 6 months before the first dose.
10. Newly diagnosed thromboembolic events requiring treatment within 6 months before the first dose.
11. Other malignant tumors diagnosed within 5 years before the first dose.
12. Known allergy to any component of KH617.
13. Positive human immunodeficiency virus (HIV) antibodies, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, and the presence of untreated or currently treated tuberculosis in the patient.
14. Patients who have received allogeneic cell or solid organ transplantation.
15. Active infection requiring systemic therapy.
16. Known history of psychotropic substance abuse, alcoholism, or drug abuse.
17. Other circumstances that the researcher deems unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
ORR | 54 weeks
PFS-6 | 54 weeks
TEAE | 54 weeks

SECONDARY OUTCOMES:
DOR | 54 weeks
PFS | 54 weeks
OS | 54 weeks
EORTC QLQ-BN20 | 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Titan Hospital,Capital Medical University